CLINICAL TRIAL: NCT03029065
Title: Detection of CSF Next Generation Sequencing in the Application of Brain Metastases From Lung Adenocarcinoma or Meningeal Metastasis
Acronym: CSF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Rongjie Tao, Shandong Cancer Hospital and Institute, Shandong Cancer Hospital and Institute
Other Study IDs: ShandongCHI004
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Recruitment
Keywords: lung Adenocarcinoma with brain (meningeal) metastasis
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Anticoagulated whole blood, anticoagulated cerebrospinal fluid and tumor tissue were collected. DNA was extracted from tumor tissues, genomic DNA was extracted from leukocytes, and cfDNA was extracted from plasma and cerebrospinal fluid.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- lung adenocarcinoma with brain (meningeal) metastasis

SUMMARY:
This study aimed to detect cell free DNA (cfDNA) in the cerebrospinal fluid and plasma, and to determine whether cfDNA can be used for concomitant diagnosis to improve the treatment efficacy and prognosis of patients with brain (meningeal) metastasis by monitoring tumor-related genetic mutations in cfDNA in the plasma and cerebrospinal fluid.

DETAILED DESCRIPTION:
This study planned to enroll 50 patients with lung cancer diagnosed with brain (meningeal) metastases, and all cases were slated to receive radiotherapy and targeted therapy. Patients' clinical data were collected (including but not limited to: age at diagnosis with brain (meningeal) metastases, KPS score, smoking history, stage of disease at diagnosis, time to progress to brain metastases, number of brain metastases, extracranial metastases (ECM), and systemic disease at the time of brain metastases. Anticoagulated whole blood and anticoagulated cerebrospinal fluid were collected before local treatment (samples of primary cancer tissue and metastatic carcinoma of some patients were preserved) and at 7 days, 1 month, 3 months, as well as 6 months after the treatment (time of sample retention was to be determined, Figure 2). DNA was extracted from tumor tissues, genomic DNA was extracted from leukocytes, and cfDNA was extracted from plasma and cerebrospinal fluid, for complete quantitative detection of DNA, DNA library construction, as well as targeted capture sequencing. Tumor-related genes were analyzed, and changes in the tumor burden during the treatment process were evaluated. The clinical significance of cfDNA in the plasma and cerebrospinal fluid for treatment efficacy and prognosis was evaluated, and compared with that of clinical indicators of treatment efficacy.

This study involved two stages. The first stage was a pre-experiment: samples were retained from 3-5 cases, and mutations in tumor-related genes in the cfDNA in plasma and cerebrospinal fluid were compared. The investigators analyzed, combined with clinical indicators, whether mutations of cfDNA in plasma accord with that of the cerebrospinal fluid and whether mutations of cfDNA in cerebrospinal can reflect the mutational status of tumor cells. The second phase was conducted by expanding the number of cases, based on the first stage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed diagnosis of lung adenocarcinoma with brain (meningeal) metastasis.
2. Samples collection should be allowed.

Exclusion Criteria:

1. Pregnant women
2. Minors (subjects less than 18 years of age)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Ages Eligible for Study: 18 Years and older (Adult, Senior) Sexes Eligible for Study: All Accepts Healthy Volunteers: No
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
investigate new diagnosis method for lung adenocarcinoma with brain (meningeal) metastasis | Participants are followed in 6 months after treatment
  Investigate whether the cfDNA can be used for concomitant diagnosis to improve the treatment efficacy and prognosis of patients with brain (meningeal) metastasis by monitoring tumor-related genetic mutations in cfDNA in the plasma and cerebrospinal fluid.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Luo N, Gao Y, Wu Y, Qin X, Qi Y, Sun T, Tao R, Qi C, Liu B, Yuan S. The joint detection of CEA and ctDNA in cerebrospinal fluid: an auxiliary tool for the diagnosis of leptomeningeal metastases in cancer. J Cancer Res Clin Oncol. 2023 May;149(5):1679-1690. doi: 10.1007/s00432-022-04053-7. Epub 2022 May 18. PMID 35583828